CLINICAL TRIAL: NCT02673463
Title: Improved Exercise Tolerance in Participants With PReserved Ejection Fraction by Spironolactone on Myocardial Fibrosis in Atrial Fibrillation
Brief Title: Spironolactone in Atrial Fibrillation
Acronym: IMPRESS-AF
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RG_14-150
Record Dates: First submitted 2016-02-01; First posted 2016-02-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Spironolactone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Spironolactone (Experimental): Spironolactone 25 mg once daily for 2 years
  Interventions: Drug: Spironolactone
- Placebo (Placebo Comparator): Matched placebo once daily for 2 years
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Spironolactone — 25 mg once daily
  Other Names: Aldactone
  Arms: Spironolactone
Drug: Placebo — Visually identical to spironolactone, once daily
  Arms: Placebo

SUMMARY:
This study aims to assess whether treatment with a drug called spironolactone, which is an aldosterone inhibitor, can improve ability to cope with exertion, quality of life and ability of the heart to relax better in symptomatic patients with atrial fibrillation with preserved pumping capacity.

DETAILED DESCRIPTION:
IMPRESS-AF study is a double-blinded randomised placebo-controlled trial of 2-year treatment with an aldosterone antagonist, spironolactone (25mg once daily) vs placebo in 250 patients with symptomatic chronic atrial fibrillation and preserved left ventricular contractility (both added to the current optimised care). The trial will establish impact of spironolactone on the primary outcome of exercise tolerance (peak oxygen consumption on cardiopulmonary exercise testing) and secondary outcomes: (i) health-related quality of life (assessed using the validated Minnesota Living with Heart Failure and EuroQol EQ-5D questionnaires self-completed by patients), and (ii) left ventricular diastolic function (E/e' ratio on echocardiography) - all assessed at baseline and at 2 years; (iii) rates of all-cause hospitalisations during 2-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Permanent AF
* Left ventricular ejection fraction >= 55% as established by echocardiography
* Able to perform cardio-pulmonary exercise testing using a cycling ergometer and complete quality of life questionnaires in English or in their native language.

Exclusion Criteria:

* Severe systemic illness (life expectancy <2 years)
* Severe chronic obstructive pulmonary disease (e.g., requiring home oxygen or chronic oral steroid therapy)
* Severe mitral/aortal valve stenosis/regurgitation
* Significant renal dysfunction (serum creatinine 220 µmol/L or above), anuria, active renal insufficiency, rapidly progressing or severe impairment of renal function, confirmed or suspected renal insufficiency in diabetic patients/ diabetic nephropathy
* Increase in potassium level to >5mmol/L
* Recent coronary artery bypass graft surgery (within 3 months)
* Use of aldosterone antagonist within 14 days before randomisation
* Use of or potassium sparing diuretic within 14 days before randomisation
* Systolic blood pressure >160 mm Hg
* Addison's disease
* Hypersensitivity to spironolactone or any of the ingredients in the product
* Any participant characteristic that may interfere with adherence to the trial protocol

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
Exercise tolerance (cardiopulmonary exercise testing) | 2 years of treatment
  Improvement in exercise tolerance (assessed using peak oxygen consumption on cardiopulmonary exercise testing)

SECONDARY OUTCOMES:
Quality of life (MLWHF) | 2 years of treatment
  Improvement in quality of life assessed using MLWHF questionnaire
Quality of life (EQ-5D) | 2 years of treatment
  Improvement in quality of life assessed using EQ-5D questionnaire
Left ventricular diastolic function | 2 years of treatment
  Improvement in diastolic function assessed using echocardiography (E/e' ratio)
Exercise tolerance (6-minute walk test) | 2 years of treatment
  Improvement in exercise tolerance (assessed using 6-minute walk test)
Rates of all-cause hospitalisations | 2 years of treatment
Spontaneous return to sinus rhythm on electrocardiogram | 2 years of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Gregory YH Lip, MD, Principal Investigator — University of Birmingham; Eduard Shantsila, PhD, Principal Investigator — University of Birmingham; Paulus Kirchhof, PhD, Principal Investigator — University of Birmingham
Locations (1):
- University of Birmingham Institute of Cardiovascular Sciences, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Shantsila E, Shahid F, Sun Y, Deeks J, Calvert M, Fisher JP, Kirchhof P, Gill PS, Lip GYH. Spironolactone in Atrial Fibrillation With Preserved Cardiac Fraction: The IMPRESS-AF Trial. J Am Heart Assoc. 2020 Sep 15;9(18):e016239. doi: 10.1161/JAHA.119.016239. Epub 2020 Sep 10. PMID 32909497
- [Derived] Shantsila E, Haynes R, Calvert M, Fisher J, Kirchhof P, Gill PS, Lip GY. IMproved exercise tolerance in patients with PReserved Ejection fraction by Spironolactone on myocardial fibrosiS in Atrial Fibrillation rationale and design of the IMPRESS-AF randomised controlled trial. BMJ Open. 2016 Oct 5;6(10):e012241. doi: 10.1136/bmjopen-2016-012241. PMID 27707827